CLINICAL TRIAL: NCT06456216
Title: Performance Evaluation of Diagnostic Accuracy (Sensitivity and Specificity) of PanTum Detect Test for Detection of Solid Tumours in Known Cancer Population (Sick Population) and in Cancer Free (Healthy) Population.
Brief Title: Performance Evaluation of Diagnostic Accuracy of PanTum Detect Test for Detection of Solid Tumours in Known Cancer Population and in Cancer Free Population.
Status: Completed | Type: Observational
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Other Study IDs: MOI-PAN-2022
Record Dates: First submitted 2024-06-05; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PanTum Detect uses the biomarkers Apo10 and TKTL1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Performance evaluation of diagnostic accuracy (Sensitivity and Specificity) of PanTum detect Test for detection of solid tumours in known cancer population (Sick population) and in cancer free (Healthy) population.

DETAILED DESCRIPTION:
PanTum Detect is a simple blood test that can detect presence of solid tumors using two important tumor biomarkers - Apo 10 and TKTL-1. Most tumors develop slowly and gradually. From the first tumor cell, to the identification of the tumor itself, there can be a timespan of many years. The turning point where a locally growing tumor develops into an invasive, metastasizing cancer is paramount for curability. It is the objective of PanTum Detect to detect a tumor in time before this critical turning point. Such locally growing tumors can often easily be removed by surgery or treated successfully

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent
2. sick population with hiostopathology proven diagnosis
3. age 30-75 years
4. newly diagnosed case of solid tumor.

Exclusion Criteria:

1. history of past surgery within 8 weeks.
2. history of any chemotherapy, vaccination etc

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: this evaluation study will be done in 3 groups of 60 subjects each using 3 differents lots of pantum detect test kit. each group will have an equal population of patients with primary tomur disease( the sick population) and healthy populations.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Performance evaluation of diagnostic accuracy (Sensitivity and Specificity) of PanTum detect Test for detection of solid tumours in known cancer population (Sick population) and in cancer free (Healthy) population. | 1 YEAR
  PanTum Detect is a simple blood test that can detect presence of solid tumors using two important tumor biomarkers - Apo 10 and TKTL-1. Most tumors develop slowly and gradually. From the first tumor cell, to the identification of the tumor itself, there can be a timespan of many years. The turning point where a locally growing tumor develops into an invasive, metastasizing cancer is paramount for curability. It is the objective of PanTum Detect to detect a tumor in time before this critical turning point. Such locally growing tumors can often easily be removed by surgery or treated successfully.

CONTACTS AND LOCATIONS:
Overall Officials: Harit Chaturvedi, MCH, Principal Investigator — Max Super Speciality Hospital, Saket
Locations (1):
- Max Super Speciality Hospital, A Unit of Devki Devi Foundation, New Delhi, India